CLINICAL TRIAL: NCT05069168
Title: Predictors of Left Ventricular Systolic Function Recovery After Transcatheter Aortic Valve
Brief Title: Predictors of Left Ventricular Systolic Function Recovery After Transcatheter Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Anwar S Helen, Principle investigator, Assiut University
Other Study IDs: TAVR
Record Dates: First submitted 2021-09-12; First posted 2021-10-06 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-02

CONDITIONS: Left Ventricular Systolic Function
MeSH Terms: interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LVEFrecovery: patient who shows improvement of left ventricular systolic function
  Interventions: Diagnostic Test: Echocardiography before and after TAVR
- Non LVEF recovery: patient who don't show improvement of left ventricular systolic function
  Interventions: Diagnostic Test: Echocardiography before and after TAVR

INTERVENTIONS:
Diagnostic Test: Echocardiography before and after TAVR — Evaluation of severity of aortic stenosis using :peak velocity ,peak and mean pressure gradient and aortic valve area by continuity equation.-Evaluation of left ventricular dimensions ,volumes and systolic function as assessed by ejection fraction (EF) by m-mode and biplane simpson's method at apical 4 and 2 chambers view Speckle tracking echocardiography(STE) Apical four-, three-, and two-chamber views were used to obtain longitudinal and circumferential strain before and follow-up after TAVR.
  cardiac CT :Routine full protocol before TAVR for evaluation and Detection and calculation of left ventricular fibrosis using extracellular volume.
  Coronary angiography:evaluate the presence of CAD and calculation of syntax score(SS)
  Other Names: cardiac computed tomography and coronary angiography

SUMMARY:
Investigate the preprocedural predictors of left ventricular systolic function Recovery after TAVR

DETAILED DESCRIPTION:
Calcific aortic stenosis (AS) is the most common valve disease in the western world requiring intervention,Although Surgical Aortic Valve Replacement (SAVR) was considered as the first therapeutic method, approximately one-third of AS patients cannot undergo SAVR due to its' high risk or contraindication.

Since Transcatheter Aortic Valve Replacement (TAVR)was performed for the first time in 2002,TAVR has emerged as a growing prevalent treatment on severe symptomatic AS with the procedure initially performed on the inoperable patients with intermediate and high risks.

Recently, the Food and Drug Administration had approved it on low-risk symptomatic subjects.

AS has to be considered a disease of the left ventricle (LV) rather than purely affecting the aortic valve, Approximately one-third of patients with severe symptomatic AS have LV systolic dysfunction .

Recovery of LV ejection fraction (LVEF) is associated with improvements in clinical outcomes after TAVR as shown by a lot of studies.

The Placement of Aortic Transcatheter Valves (PARTNER) trial demonstrated that recovery of LV function in patients with severe symptomatic AS and LV systolic dysfunction who underwent TAVR, occurs in 40% to 50% of patients .

Higher trans-aortic mean pressure gradient , less LV hypertrophy, Less LV fibrosis and absence of AF are predictors of recovery of LV function after TAVR .

However, there is still a scanty data about the predictors of LV function recovery after TAVR.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic severe aortic stenosis eligible for TAVR with LV systolic function less than 50%.

Exclusion Criteria:

* Severe Rheumatic or degenerative mitral regurgitation.
* Previous Valve Replacement.
* Previous myocardial infarction.
* Previous Coronary Artery By Bass Graft (CABG)Surgery.
* Post TAVR significant paravalvular leakage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with symptomatic severe aortic stenosis eligible for TAVR with LV systolic function less than 50%
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
left ventricular systolic function recovery by ejection fraction | 30 days post TAVR
  absolute increase of ≥10% in EF compared with baseline
left ventricular systolic function recovery by STE | 30 days post TAVR
  Myocardial recovery by STE is defined as a ≥20% relative increase in the magnitude of global longitudinal strain compared with baseline

SECONDARY OUTCOMES:
Quality of life assessment | 30days post TAVR
  NIHA class .

CONTACTS AND LOCATIONS:
Overall Officials: Hatem A Helmy, Study Director — Assiut University
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Passeri JJ, Elmariah S, Xu K, Inglessis I, Baker JN, Alu M, Kodali S, Leon MB, Svensson LG, Pibarot P, Fearon WF, Kirtane AJ, Vlahakes GJ, Palacios IF, Douglas PS; PARTNER Investigators. Transcatheter aortic valve replacement and standard therapy in inoperable patients with aortic stenosis and low EF. Heart. 2015 Mar;101(6):463-71. doi: 10.1136/heartjnl-2014-306737. Epub 2015 Jan 13. PMID 25586156
- [Background] Sato K, Kumar A, Jones BM, Mick SL, Krishnaswamy A, Grimm RA, Desai MY, Griffin BP, Rodriguez LL, Kapadia SR, Obuchowski NA, Popovic ZB. Reversibility of Cardiac Function Predicts Outcome After Transcatheter Aortic Valve Replacement in Patients With Severe Aortic Stenosis. J Am Heart Assoc. 2017 Jul 11;6(7):e005798. doi: 10.1161/JAHA.117.005798. PMID 28698259
- [Background] Han D, Tamarappoo B, Klein E, Tyler J, Chakravarty T, Otaki Y, Miller R, Eisenberg E, Park R, Singh S, Shiota T, Siegel R, Stegic J, Salseth T, Cheng W, Dey D, Thomson L, Berman D, Makkar R, Friedman J. Computed tomography angiography-derived extracellular volume fraction predicts early recovery of left ventricular systolic function after transcatheter aortic valve replacement. Eur Heart J Cardiovasc Imaging. 2021 Jan 22;22(2):179-185. doi: 10.1093/ehjci/jeaa310. PMID 33324979
- [Background] Jeong YJ, Ahn JM, Kang DY, Park H, Ko E, Kim HJ, Kim JB, Choo SJ, Lee SA, Park SJ, Kim DH, Park DW. Incidence, Predictors, and Prognostic Impact of Immediate Improvement in Left Ventricular Systolic Function After Transcatheter Aortic Valve Implantation. Am J Cardiol. 2021 Aug 1;152:99-105. doi: 10.1016/j.amjcard.2021.04.037. Epub 2021 Jun 11. PMID 34127247